CLINICAL TRIAL: NCT05492331
Title: A Randomized Controlled Trial to Assess the Effect of Music Therapy on the Anxiety of Patients Undergoing Intrauterine Insemination
Brief Title: A Study of Music Therapy to Support Intrauterine Insemination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Alessandra (Ali) J. Ainsworth, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-006147
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Intrauterine Insemination
Keywords: Music Therapy
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy during the IUI procedure (Experimental): Subjects undergoing an intrauterine insemination (IUI) procedure will experience music therapy during the procedure.
  Interventions: Other: Music Therapy
- Standard of Care (No Intervention): Subjects will receive standard of care for intrauterine insemination (IUI) procedure.

INTERVENTIONS:
Other: Music Therapy — Patient preferred artist or music genre to be playing from an iPad
  Arms: Music Therapy during the IUI procedure

SUMMARY:
The purpose of this research is to learn if playing music in the room during an intrauterine insemination procedure decreases anxiety and pain for patients at the time of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* IUI must be performed in the Reproductive Endocrinology and Infertility offices at Mayo Clinic in Rochester.
* IUI procedure must be on a weekday.
* IUI procedure is scheduled to be completed by a nurse in the REI Department.

Exclusion Criteria:

* Not English speaking.
* IUI procedure on a weekend day.
* IUI procedure is scheduled with an MD provider (known or expected to be difficult).
* Planned IUI procedure is cancelled prior to undergoing the procedure.
* The patient has a documented diagnosis of complete hearing loss or significant hearing impairment in both ears.
* The patient has previous participated or declined enrollment in the study during a prior IUI procedure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Change in anxiety | Baseline, during IUI procedure (approximately 20 minutes), after IUI procedure (approximately 5 minutes)
  Assessed using the 100-mm Visual Analogue Scale (VAS). The VAS line will be 100 mm long with no intermediate delineations. Each end will be marked with "No anxiety" on the left, and "Worst anxiety" on the right. Participants will identify their anxiety level by indicating a point on the line between each end. That point will be measured from the "No anxiety" end, and the number of millimeters will be reported as the pain score.

SECONDARY OUTCOMES:
Change in pain score | Baseline, during IUI procedure (approximately 20 minutes), after IUI procedure (approximately 5 minutes)
  Assessed using the Wong Baker Pain Rating. Subjects will place a mark on the face that best describes their pain level. Uses a 0-10 scale, where 0 represents "No pain" on the left, and 10 represents "Worst possible pain" on the right.
Pregnancy rate | 1 year
  Number of subjects to become pregnant

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ainsworth, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baumgarten SC, Chen V, Ogle AJ, Fought AJ, Li Y, Ainsworth AJ. Effect of music on anxiety during intrauterine insemination: a randomized controlled trial. F S Rep. 2025 May 22;6(3):381-387. doi: 10.1016/j.xfre.2025.05.008. eCollection 2025 Sep. PMID 41054719
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials